CLINICAL TRIAL: NCT03316027
Title: Adherence Rate to Disease Modifying Anti Rheumatic Drugs in Egyptian Patients With Rheumatoid Arthritis: Possible Predictions and Correlations
Brief Title: Adherence Rate to DMARDS in Egyptian Patients With RA
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Esraa Moustafa Mohammed, Principal investigator, Assiut University
Other Study IDs: DMARDS in RA
Record Dates: First submitted 2017-09-30; First posted 2017-10-20 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study aims at determining adherence rate to DMARDS and predicting factors affecting treatment adherence among sample of Egyptian patients with RA.

DETAILED DESCRIPTION:
Rheumatoid arthritis (RA) is an autoimmune disease that causes inflammation of the joints. It is chronic disease and often progressive in course and has a strong impact on people's everyday lives.

Disease Modifying Anti-Rheumatic Drugs (DMARDS), such as methotrexate, leflunomide, hydroxychloroquine, and sulfasalazine are the cornerstone of therapy in RA and are invariably used as initial therapy.

These drugs have shown to retard disease progression including joint destruction.

It is believed that adherence to treatment is crucial for successful therapy, however, non-adherence is a substantial problem in patients with chronic rheumatic conditions, including RA.

Previous studies have reported that DMARDS non adherence results in more disease activity, loss of function, and a lower quality of life.

The depression is a common co-morbidity in RA, its presence can alter the course of RA negatively via cognitive-behavioral or inflammatory pathways: patients with concurrent depression suffer from more pain, show a heightened disease activity.

As non-adherence to medication regimen is considered a serious public health issue that can have great impact on clinical and economic consequences. therefore, it is crucial for health care providers to assess the patient condition, predict the possible causes of non-adherence, and put a policy for increasing medication adherence and achieving the best health outcome.

Also, improving medication adherence enhances patients' safety and health condition.

ELIGIBILITY:
Inclusion Criteria:

1. Age more than or equal 18 years old.
2. On current diagnosis of RA determined by a Rheumatologist according to 2010 ACR/EULAR classification criteria for RA.
3. On current treatment with one or more of DMARDS from at least 6 months duration.
4. Patients with cognitive level enabling them to interact in the study. -

Exclusion Criteria:

1. Age less than 18 years old.
2. Patients receiving one or more of DMARDS of period less than 6 months.
3. Patients with psychiatric diagnosis other than effective disorder.
4. Patients with associated disability due to neurological disorder or trauma.
5. Patients with major internal organ failure e.g. heart failure, end stage renal disease or hepatic failure.
6. Patients with severe cognitive impairment interfering with the proper communication and interaction within the study process.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients from both sex, aged more than or equal 18 years old, attending Physical Medicine, Rheumatology and Rehabilitation department, Assiut University Hospital, on current diagnosis of RA from at least 6 months and current treatment with one or more of DMARDS, with cognitive level enabling them to interact in the study, and free from psychiatric diagnosis other than effective disorder, associated disability due to neurological disorder or trauma and also free from major internal organ failure.
Sampling Method: Non-Probability Sample
Enrollment: 73 (Estimated)
Dates: Start 2019-11 (Estimated); Primary Completion 2019-11 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients adherent to the treatment through MMAS-8. | 6 months.
  The use of Morisky Medication Adherence Scale 8- item (MMAS-8) to determining percentage of patients adherent to treatment.

REFERENCES:
- [Background] Harrold LR, Andrade SE. Medication adherence of patients with selected rheumatic conditions: a systematic review of the literature. Semin Arthritis Rheum. 2009 Apr;38(5):396-402. doi: 10.1016/j.semarthrit.2008.01.011. Epub 2008 Mar 12. PMID 18336875
- [Background] Contreras-Yanez I, Ponce De Leon S, Cabiedes J, Rull-Gabayet M, Pascual-Ramos V. Inadequate therapy behavior is associated to disease flares in patients with rheumatoid arthritis who have achieved remission with disease-modifying antirheumatic drugs. Am J Med Sci. 2010 Oct;340(4):282-90. doi: 10.1097/MAJ.0b013e3181e8bcb0. PMID 20881757
- [Background] Wells G, Becker JC, Teng J, Dougados M, Schiff M, Smolen J, Aletaha D, van Riel PL. Validation of the 28-joint Disease Activity Score (DAS28) and European League Against Rheumatism response criteria based on C-reactive protein against disease progression in patients with rheumatoid arthritis, and comparison with the DAS28 based on erythrocyte sedimentation rate. Ann Rheum Dis. 2009 Jun;68(6):954-60. doi: 10.1136/ard.2007.084459. Epub 2008 May 19. PMID 18490431
- [Background] Bruce B, Fries JF. The Stanford Health Assessment Questionnaire: a review of its history, issues, progress, and documentation. J Rheumatol. 2003 Jan;30(1):167-78. PMID 12508408
- [Background] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820